CLINICAL TRIAL: NCT06547593
Title: A Multifaceted Nutrition Intervention for Frailty in the Community Elderly: a Randomized Controlled Trial
Brief Title: A Multifaceted Nutrition Intervention for Frailty in the Community Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhaofeng Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhaofeng Zhang, Associate Professor, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MINUTE
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Frail; Elderly; Nutrition Disorders in Old Age
Keywords: multifaceted nutrition; frail; elderly; community
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutritional Intervention Group (Experimental): In this group, based on routine health management, a 3-month multifaceted nutrition intervention and a 9-month follow-up will be conducted. The specific content is as follows:
  1. Anti-inflammatory dietary management: the elderly will receive an anti-inflammatory dietary menu designed based on the Chinese Dietary Guidelines for the Elderly (2022 Edition) provided by researchers.
  2. Personalized nutritional intervention management: To ensure the compliance and participation of the elderly, a variety of health intervention materials will be provided. WeChat groups will be established to record the dietary status of the research subjects.
  3. Health education: Nutrition and health knowledge lecture will be held for elderly family caregivers and the elderly themselves every two weeks.
  Interventions: Behavioral: multifaceted nutrition intervention
- Nutritional and Exercise Combined Intervention Group (Experimental): To investigate the combined effects of nutrition and exercise, this group added exercise intervention in addition to the corresponding intervention measures of the nutrition intervention group. The subjects were required to exercise 3 times a week, 1 hour each time. The project included 10 minutes of warm-up exercises (stretching), 10-20 minutes of aerobic exercise (balance ability, leg and core muscle strength, etc.), 10-20 minutes of muscle resistance strength training (legs, buttocks, feet, upper limbs, etc.) and 10 minutes of relaxation training. All exercise programs were uniformly trained by professional coaches, and compliance was ensured by uploading photos to punch the clock. The intervention period is 3 months, with a follow-up of 9 months.
  Interventions: Behavioral: Nutritional and Exercise Combined Intervention
- Control Group (Placebo Comparator): The control group will undergo routine community health management, including regular chronic disease health education lectures, provision of health education materials, health counseling services, and comprehensive health examinations by qualified medical professionals.
  At the beginning and end of the intervention, as well as at a 9-month follow-up, the study subjects were evaluated to understand the sustainability of the intervention after the project was completed, and to explore the management mode of sustainable intervention.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: multifaceted nutrition intervention — In this group, a 3-month multifaceted nutrition intervention will be conducted. The specific content is as follows:
  1. Anti-inflammatory dietary management: the elderly will receive an anti-inflammatory dietary menu designed based on the Chinese Dietary Guidelines for the Elderly (2022 Edition) provided by researchers.
  2. Personalized nutritional intervention management: WeChat groups will be established to record the dietary status of the research subjects. The research subjects will be asked to keep a dietary diary and take photos of their diet daily. Trained researchers will record their daily diet and provide timely feedback to the research subjects.
  3. Health education: Nutrition and health knowledge lecture will be held for elderly family caregivers and the elderly themselves every two weeks. The content will include basic knowledge of frailty, prevention and treatment guidance, health outcomes, medication management, and healthy behaviors.
  Arms: Nutritional Intervention Group
Behavioral: Nutritional and Exercise Combined Intervention — To investigate the combined effects of nutrition and exercise, this group added exercise intervention in addition to the corresponding intervention measures of the nutrition intervention group. The subjects were required to exercise 3 times a week, 1 hour each time. The project included 10 minutes of warm-up exercises (stretching), 10-20 minutes of aerobic exercise (balance ability, leg and core muscle strength, etc.), 10-20 minutes of muscle resistance strength training (legs, buttocks, feet, upper limbs, etc.) and 10 minutes of relaxation training. All exercise programs were uniformly trained by professional coaches, and compliance was ensured by uploading photos to punch the clock. The intervention period is 3 months, with a follow-up of 9 months.
  Arms: Nutritional and Exercise Combined Intervention Group
Behavioral: Control Group — The control group will undergo routine community health management, including regular chronic disease health education lectures, provision of health education materials, health counseling services, and comprehensive health examinations by qualified medical professionals.
  Arms: Control Group

SUMMARY:
With world's older population is rapidly increasing. China's population aging process is also accelerating. Studies have shown that persistent frailty can increase the incidence of negative events in the elderly. However, research on elderly frailty in China is still in its early stages, and existing research in China mainly focuses on the definition of frailty, evaluation tools for frailty, and cross-sectional surveys of small populations. There is currently limited research on interventions.

The MultIfaceted NUtrition inTErvention for Frailty (minute) trial is a randomized, controlled trial to explore the trajectory characteristics and influencing factors of frailty in the community, the impact of nutritional interventions on the developmental trajectory of frailty in the elderly in the community and the management model and appropriate technology for the sustainable intervention of frailty in the elderly based on the community.

A total of 315 frail older adults will be recruited from Beijing. After the screening period, the compliant participants will be randomized to the control group, the nutrition intervention group with the nutrition intervention alone, or the combined nutrition intervention group with combining exercise and nutrition, on a 1:1:1 ratio, for 3 months. The primary outcome is the change in SPPB from the baseline to the end of the study. The change in SPPB as a primary outcome, and frailty status, demographic information, health status, nutrition assessment, comprehensive geriatric assessment status, quality of life, intrinsic capacity, and mental elasticity as secondary outcomes will be measured using validated questionnaires and clinical examinations.

This trial adheres to the Declaration of Helsinki and guidelines of Good Clinical Practice. Signed informed consent will be obtained from all participants. The trial has been approved by the Peking University Institutional Review Board (approval number: IRB00001052-23178). The results will be disseminated through academic conferences and publications in international peer-reviewed journals.

DETAILED DESCRIPTION:
The global elderly population is rapidly increasing, with the 65-and-over age group being the fastest growing. Currently, about 9% of the world's population is over 65, and this proportion is projected to reach 16% by 2050. The silvering of China's population continues its steady march. By the end of 2023, the population aged 60 and above is 296.97 million, accounting for 21.1% of the national population, of which 216.76 million are aged 65 and above, accounting for 15.4% of the national population. As China's population continues to age, the silver tsunami shows no signs of abating. By 2030, it is estimated that the number of elderly individuals aged 65 and above will have surged to approximately 240 million. And by 2050, the ranks of octogenarians and above are projected to reach a staggering 100 million. The overall health status of China's elderly population is a cause for concern. More than 80% of individuals aged 65 and above suffer from at least one chronic disease, and by the age of 75, this number increases to at least three. Approximately 44 million elderly citizens are either partially or fully disabled, casting a long shadow over their own lives, placing a significant burden on their families, and society. The health of China's elderly has become a pressing public health issue that demands the attention of the entire nation. Frailty is a geriatric syndrome characterized by an increased vulnerability to stressors. It is a state of diminished physiological reserve and impaired function across multiple organ systems, leading to increased dependency and mortality. Epidemiological data suggest that the prevalence of frailty in the elderly population ranges from approximately 4.9% to 27.3%. Among community-dwelling elderly individuals, the prevalence is estimated to be between 6.9% and 14.9%. The incidence of frailty increases with advancing age, with over 25% of individuals aged 85 and older experiencing this debilitating condition. Research has painted a sobering picture of the consequences of persistent frailty in the elderly population. It has been shown to increase the risk of a cascade of negative events, including falls, disability, delirium, hospitalization, and even premature mortality. The risk of morbidity and mortality escalates significantly, with a 68% increase in all-cause mortality for every 0.1-unit increase in the frailty index (HR=1.68, 95% CI: 1.66-1.71). Frailty also places a heavy burden on caregivers and healthcare systems, straining resources and exacerbating the challenges of caring for an aging population. Furthermore, frail elderly individuals are particularly vulnerable to precipitous declines in health, even from minor stressors such as infections, new medications, falls, constipation, or urinary retention. These events can trigger a downward spiral, leading to hospitalization, disability, and even death, severely compromising the quality of life for elderly individuals and placing a greater demand on healthcare services. In the global tapestry of frailty research, interventions have largely focused on isolated threads, such as exercise regimens, nutritional counseling, risk factor modification, and comprehensive care. However, the intricate web of frailty demands a more holistic approach, one that weaves together these diverse strands. There is a notable lack of research investigating comprehensive intervention measures. It is of utmost importance to conduct community-based research to explore a comprehensive nutritional intervention model for frailty that is tailored to the unique characteristics of the Chinese population, scientifically sound, and sustainable.

ELIGIBILITY:
Inclusion Criteria:

1. Frailty assessed by the frail phenotype
2. Aged between 65 and 85 years old

Exclusion Criteria:

1. Multiple serious diseases such as stroke, cerebral infarction, tumors, and severe cardiovascular and cerebrovascular diseases
2. Disability, dementia; severe visual and hearing impairments, and physical activity impairment
3. Moderate to severe anxiety and depression
4. Unable to complete this study as requested

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) score | at the 3-month intervention and at the 3-month, 6-monthand 12-month follow-up investigations
  The primary outcome was the change in the Short Physical Performance Battery (SPPB) score between groups, and the change from baseline to the end of the study.
frailty scores | at the 3-month intervention and at the 3-month, 6-month and 12-month follow-up investigations
  The frailty scores were evaluated using Fried Frailty Phenotype and Tilburg Frailty Indicator

SECONDARY OUTCOMES:
frailty trajectories | at the 3-month intervention and at the 3-month, 6-month and 12-month follow-up investigations
  Changes in frailty trajectories before and after the intervention, as measured by the Frailty Index.
intrinsic capacity | at the 3-month intervention and at the 3-month, 6-month and 12-month follow-up investigations
  Changes in intrinsic capacity before and after the intervention, and between groups; The intrinsic capacity is measured using the World Health Organization's (WHO) Integrated Care for Older People (ICOPE) approach.
Malnutrition risk assessment | at the 3-month intervention and at the 3-month, 6-month and 12-month follow-up investigations
  Measured by 《Malnutrition Risk Assessment Form for the Elderly》
frailty recovery rates | at the 3-month intervention and at the 3-month, 6-month and 12-month follow-up investigations
  Difference in frailty scores before and after intervention
Serum protein | at the 3-month intervention and at the 3-month and 12-month follow-up investigations
  serum total protein, albumin and transferrin
Urine 8-hydroxyguanosine (8-oxo-Gsn) | at the 3-month intervention and at the 3-month and 12-month follow-up investigations
  Urine oxidation marker 8-hydroxyguanosine (8-oxo-Gsn) level
Serum inflammatory factors | at the 3-month intervention and at the 3-month and 12-month follow-up investigations
  C-reactive protein (CRP), interleukin-6 (IL-6), tumor necrosis factor - α (TNF - α), insulin-like growth factor-1 (IGF-1), C-X-C-motif chemokine 10 (CXCL10), chemokine C-X3-C-based ligand 1 (CX3CL1) in serum using ELISA
changes in serum differential metabolites | At the beginning of the intervention and in the third month of the intervention
  Using non targeted metabolomics methods to examine the changes in serum differential metabolites in each group before and after intervention, and elucidate the mechanism of intervention
changes in gut microbiota | At the beginning of the intervention and in the third month of the intervention
  Using 16S sequencing method to detect changes in gut microbiota and differential bacterial genera among groups
participants' satisfaction | At the beginning of the intervention and in the third month of the intervention
  participants satisfaction and acceptability is evaluated using a self-made scale
cognition function | at the 3-month intervention and at the 6-month and 12-month follow-up investigations
  cognition function is evaluated using Mini-Mental State Examination, MMSE
Sleep conditions | at the 3-month intervention and at the 6-month and 12-month follow-up investigations
  Sleep conditions is evaluated using Pittsburgh sleep quality index
adverse event | at the 3-month intervention and at the 6-month and 12-month follow-up investigations
  serious adverse events, unexpected adverse events, and adverse events that occurred while the participant was under the supervision or guidance of study staff either onsite or offsite.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaofeng Zhang, Doctor, Principal Investigator — Peking University
Locations (1):
- Qingta Community Health Service Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Han Y, Zhang H, Sun M, Ma Y, Tu Y, Tian J, Fan R, Zhu W, Zhang Z. Multifaceted Nutrition Intervention for Frail Elderly in the Community: Protocol of a Randomized Controlled Trial (The MINUTE Study). Nutrients. 2025 Oct 13;17(20):3213. doi: 10.3390/nu17203213. PMID 41156465